CLINICAL TRIAL: NCT00940862
Title: Pilot Study on the Effect of Adalimumab on Vascular Inflammation in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: Effect of Adalimumab on Vascular Inflammation in Patients With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovaderm Research Inc. (Other)
Collaborators: Abbott (Industry); Montreal Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Inno-6009
Record Dates: First submitted 2009-06-22; First posted 2009-07-16 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-10

CONDITIONS: Psoriasis; Vascular Inflammation; Coronary Atherosclerosis
Keywords: psoriasis; vascular inflammation; coronary atherosclerosis
MeSH Terms: conditions — Psoriasis; Coronary Artery Disease | interventions — Adalimumab; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- adalimumab (Experimental): A total of 20 patients will be randomized to adalimumab (80 mg followed by 40 mg at week 1 and 40 mg EOW thereafter for 15 weeks)
  Interventions: Biological: adalimumab
- Non-systemic treatment. (Active Comparator): A total of 10 patients will be randomized to non systemic therapy for psoriasis (topical treatments and/or UVB phototherapy).
  Interventions: Device: UVB Phototherapy; Other: Topical treatment

INTERVENTIONS:
Biological: adalimumab — Injection of adalimumab (80 mg followed by 40 mg at week 1 and 40 mg EOW thereafter for 15 weeks)
  Other Names: Humira
  Arms: adalimumab
Device: UVB Phototherapy — This intervention can be applied alone or in combination with topical treatment. It will be performed between Day 0 and Day 112. The investigator is free to introduce or modify the topical and/or UVB regimens at any time after screening.
  Other Names: Ultra violet light B
  Arms: Non-systemic treatment.
Other: Topical treatment — This intervention can be applied alone or in combination with UVB phototherapy. It will be performed between Day 0 and Day 112. The investigator is free to introduce or modify the topical and/or UVB regimens at any time after screening. The investigator will prescribe to patients randomized in this arm a select topical product from the list:
  Calcipotriol, Calcipotriene, Dovonex, Tazorac, Tazarotene Anthralin, Corticosteroids.
  Arms: Non-systemic treatment.

SUMMARY:
This study is to determine the effect of adalimumab on inflammation of blood vessels that could lead to heart attack in patients with psoriasis. Changes to the carotid artery and ascending aorta will be evaluated in patients treated with adalimumab (systemic treatment) and compared against patients treated with a topical treatment that does not affect the entire body.

DETAILED DESCRIPTION:
Psoriasis and rheumatoid arthritis (RA) have been shown to be independent risk factors for myocardial infarction (MI). The risk is believed to be related in part to systemic inflammation associated with these diseases. Some studies have suggested that treatment of RA patients with anti-TNF alpha can decrease the risks of MI. However, we do not have data on the effect of anti-TNF alpha on coronary atherosclerosis. Adalimumab is probably the best anti-TNF alpha candidate to study for an effect on coronary atherosclerosis as it has more affinity for membrane bound TNF alpha than other anti-TNF alpha products such as etanercept and a higher global anti-TNF alpha activity in psoriasis patients.

This study involves a comparison of adalimumab administered sub-cutaneously with a loading dose of 80 mg followed by 40 mg at week 1 and 40 mg every other week thereafter for a total of 10 injections (two 40 mg injections at week 0 for a total dose of 80 mg, followed by single injections at weeks 1, 3, 5, 7, 9, 11, 13 and 15) with non systemic treatments for psoriasis (topical therapy and/or UVB therapy). Patients will be randomized (2:1) to either adalimumab or topical and/or UVB therapy for psoriasis.

If this pilot study shows that adalimumab reduces vascular inflammation in patients with psoriasis, a larger study could be undertaken to study the effect of adalimumab on coronary atherosclerotic plaques.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old and capable of giving informed consent.
* at least a 6-month history of chronic moderate to severe psoriasis and a candidate for systemic therapy.
* BSA covered with psoriasis of at least 5 % or more at Baseline.
* An history of coronary atherosclerosis or at least three risk factors among the following: hypertension, active smoking, diabetes mellitus, dyslipidemia, obesity, microalbuminuria, age above 55 years, and first degree relative with coronary atherosclerosis before 65 years.
* Patient must be on a stable dose for at least 8 weeks before baseline if taking medications used to control angina, hypertension, serum lipids and any medication that can have an effect on inflammation.
* Patient has a carotid or ascending aorta atherosclerotic plaque inflammation target-to background ratio of 1.6 or more as determined by 18-FDG uptake measured by PET scanning.
* Female patient is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile, or is of childbearing potential and practicing one of the following methods of birth control throughout the study and for 150 days after study completion:

  * condoms, sponge, foams, jellies, diaphragm or IUD.
  * contraceptives for three months prior to study drug administration
  * a vasectomized partner.
* Female patient of childbearing potential must have a negative serum pregnancy test at the Screening visit.
* Patient is judged to be in good general health as determined by the principal investigator.
* Patient will be evaluated for latent TB infection with a PPD or a Quantiferon Gold test and CXR. Patient who demonstrates evidence of latent TB infection will only be allowed to participate in the study if they are willing to use TB prophylaxis according to Canadian guidelines
* Patient must be able and willing to provide written informed consent and comply with the requirements of this study protocol.
* Patient must be able and willing to self-administer SC injections or have a qualified person available to administer SC injections.

Exclusion Criteria:

* Patient has other active skin diseases or skin infections (that may interfere with evaluation of psoriasis or with patient's safety.
* Patient has a history of an allergic reaction or significant sensitivity to constituents of study drug, including latex.
* Patient used any non-biological systemic therapy for the treatment of psoriasis less than 30 days before Day 0. Investigational chemical agents must be discontinued at least 30 days or five half-lives prior to the Baseline visit (whichever is longer).
* Patient who has used any biological therapy for the treatment of psoriasis less than 3 months (90 days) before Day 0.
* Patient is taking or requires oral or injectable corticosteroids during the study. Inhaled corticosteroids for stable medical conditions are allowed.
* Patient has used any topical treatment for psoriasis or has used phototherapy within the last 2 weeks prior to baseline (at the exception of low strength (hydrocortisone and desonide) topical corticosteroid for the face, groin (including genitals) and inframammary areas).
* Patient has received Anakinra/Kineret within the last 2 weeks prior to the Baseline visit or is likely to receive Anakinra/Kineret during the course of the study.
* Patient has a poorly controlled medical condition, such as uncontrolled diabetes, documented history of recurrent infections, unstable ischemic heart disease, congestive heart failure a left ventricular ejection fraction of less than 40%, recent stroke, chronic leg ulcer or any other condition which, in the opinion of the investigator, would put the patient at risk if participating in the study.
* Patient had a myocardial infarction or hospitalization for a cardiac condition within the past 12 weeks.
* Patient has a history of acute coronary syndrome, percutaneous coronary intervention, coronary artery bypass graft, or carotid revascularization within 12 weeks of baseline.
* Patient for whom a change in medical treatment for angina, serum lipids, hypertension or any other medication that can have a significant effect on inflammation is planned for the duration of the study.
* Patient has a history of neurologic symptoms suggestive of central nervous system demyelinating disease.
* Patient has history of cancer or lymphoproliferative disease other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix.
* Patient has a history of listeriosis, treated or untreated TB, persistent chronic infections, or recent active infections requiring hospitalization or treatment with intravenous anti-infectives within 30 days or oral anti-infectives within 14 days prior to the Baseline visit.
* Patient has received any live attenuated vaccine 28 days or less before baseline.
* Patient with hepatitis B or hepatitis C viral infection.
* Patient with any of the following: hemoglobin = 10 g/L, white blood cell count = 3.0 X 109/L, platelet count =130 X 109/L, ALT = 2 times the upper limit of normal, AST = 2 times the upper normal limit, total bilirubin = 2 times the upper normal limit or creatinine = 150 umol/L.
* Patient is currently using or plans to use anti-retroviral therapy at any time during the study.
* Patient is known to have immune deficiency or is immunocompromised.
* Female patient who is pregnant or breast-feeding or considering becoming pregnant during the study or for 150 days after the last dose of study medication.
* Patient has a history of clinically significant drug or alcohol abuse in the last year.
* Patient is considered by the investigator, for any reason, to be an unsuitable candidate for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The changes in the target (atherosclerotic plaque) to background (blood) ratio (TBR) from the carotid artery and ascending aorta in patients randomized to adalimumab as compared to patients randomized to standard non-systemic therapy. | Day -10 to -1, Day 105

SECONDARY OUTCOMES:
The changes in the TBR from a coronary artery from Day 0 to Day 105 in patients randomized to adalimumab as compared to patients randomized to standard therapy. | Day -10 to -1, Day 105.
To study changes in hs C-Reactive protein levels and serum lipids levels between Day 0 and Day 112 in patients randomized to adalimumab compared to patients randomized to standard therapy. | Day 0, 28, 56, 112
To study the safety of adalimumab in patients with psoriasis and history of coronary atherosclerosis or with at least three risk factors for coronary atherosclerosis. atherosclerosis or with at least three risk factors for coronary atherosclerosis | Day 0, 28, 56, 112, 175
To study the efficacy of adalimumab in patients with psoriasis and coronary atherosclerosis or at least three risk factors. PASI will be recorded and the percentage of patients achieving PASI 75 at Day 112 will be calculated for all patients randomized. | Day 0, 28, 56, 112

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, Principal Investigator — Innovaderm Research; Jean-Claude Tardif, MD, FRCPC, Principal Investigator — Montreal Heart Institute
Locations (2):
- Canada (2):
  - Montreal Heart Institute, Montreal, Quebec
  - Innovaderm Research Inc, Montreal, Quebec

REFERENCES:
- [Background] Choi J, Koo JY. Quality of life issues in psoriasis. J Am Acad Dermatol. 2003 Aug;49(2 Suppl):S57-61. doi: 10.1016/s0190-9622(03)01136-8. PMID 12894127
- [Background] Gelfand JM, Feldman SR, Stern RS, Thomas J, Rolstad T, Margolis DJ. Determinants of quality of life in patients with psoriasis: a study from the US population. J Am Acad Dermatol. 2004 Nov;51(5):704-8. doi: 10.1016/j.jaad.2004.04.014. PMID 15523347
- [Background] Weiss SC, Kimball AB, Liewehr DJ, Blauvelt A, Turner ML, Emanuel EJ. Quantifying the harmful effect of psoriasis on health-related quality of life. J Am Acad Dermatol. 2002 Oct;47(4):512-8. doi: 10.1067/mjd.2002.122755. PMID 12271293
- [Background] Tremblay JF, Bissonnette R. Topical agents for the treatment of psoriasis, past, present and future. J Cutan Med Surg. 2002 May-Jun;6(3 Suppl):8-11. doi: 10.1177/12034754020060S303. Epub 2002 Apr 30. No abstract available. PMID 11976984
- [Background] Guenther L, Langley RG, Shear NH, Bissonnette R, Ho V, Lynde C, Murray E, Papp K, Poulin Y, Zip C. Integrating biologic agents into management of moderate-to-severe psoriasis: a consensus of the Canadian Psoriasis Expert Panel. February 27, 2004. J Cutan Med Surg. 2004 Sep-Oct;8(5):321-37. doi: 10.1007/s10227-005-0035-1. PMID 15868311
- [Background] Langley RG, Ho V, Lynde C, Papp KA, Poulin Y, Shear N, Toole J, Zip C. Recommendations for incorporating biologicals into management of moderate to severe plaque psoriasis: individualized patient approaches. J Cutan Med Surg. 2006;9 Suppl 1:18-25. doi: 10.1007/s10227-006-0103-1. PMID 16633860
- [Background] Gelfand JM, Neimann AL, Shin DB, Wang X, Margolis DJ, Troxel AB. Risk of myocardial infarction in patients with psoriasis. JAMA. 2006 Oct 11;296(14):1735-41. doi: 10.1001/jama.296.14.1735. PMID 17032986
- [Background] Goodson N, Marks J, Lunt M, Symmons D. Cardiovascular admissions and mortality in an inception cohort of patients with rheumatoid arthritis with onset in the 1980s and 1990s. Ann Rheum Dis. 2005 Nov;64(11):1595-601. doi: 10.1136/ard.2004.034777. Epub 2005 Apr 20. PMID 15843450
- [Background] Maradit-Kremers H, Crowson CS, Nicola PJ, Ballman KV, Roger VL, Jacobsen SJ, Gabriel SE. Increased unrecognized coronary heart disease and sudden deaths in rheumatoid arthritis: a population-based cohort study. Arthritis Rheum. 2005 Feb;52(2):402-11. doi: 10.1002/art.20853. PMID 15693010
- [Background] Watson DJ, Rhodes T, Guess HA. All-cause mortality and vascular events among patients with rheumatoid arthritis, osteoarthritis, or no arthritis in the UK General Practice Research Database. J Rheumatol. 2003 Jun;30(6):1196-202. PMID 12784389
- [Background] van Leuven SI, Franssen R, Kastelein JJ, Levi M, Stroes ES, Tak PP. Systemic inflammation as a risk factor for atherothrombosis. Rheumatology (Oxford). 2008 Jan;47(1):3-7. doi: 10.1093/rheumatology/kem202. Epub 2007 Aug 16. PMID 17702769
- [Background] Moubayed SP, Heinonen TM, Tardif JC. Anti-inflammatory drugs and atherosclerosis. Curr Opin Lipidol. 2007 Dec;18(6):638-44. doi: 10.1097/MOL.0b013e3282f0ee11. PMID 17993809
- [Background] Dixon WG, Symmons DP. What effects might anti-TNFalpha treatment be expected to have on cardiovascular morbidity and mortality in rheumatoid arthritis? A review of the role of TNFalpha in cardiovascular pathophysiology. Ann Rheum Dis. 2007 Sep;66(9):1132-6. doi: 10.1136/ard.2006.063867. Epub 2007 Jan 24. PMID 17251223
- [Background] Dixon WG, Watson KD, Lunt M, Hyrich KL; British Society for Rheumatology Biologics Register Control Centre Consortium; Silman AJ, Symmons DP; British Society for Rheumatology Biologics Register. Reduction in the incidence of myocardial infarction in patients with rheumatoid arthritis who respond to anti-tumor necrosis factor alpha therapy: results from the British Society for Rheumatology Biologics Register. Arthritis Rheum. 2007 Sep;56(9):2905-12. doi: 10.1002/art.22809. PMID 17763428
- [Background] Jacobsson LT, Turesson C, Gulfe A, Kapetanovic MC, Petersson IF, Saxne T, Geborek P. Treatment with tumor necrosis factor blockers is associated with a lower incidence of first cardiovascular events in patients with rheumatoid arthritis. J Rheumatol. 2005 Jul;32(7):1213-8. PMID 15996054
- [Background] Leonardi CL, Powers JL, Matheson RT, Goffe BS, Zitnik R, Wang A, Gottlieb AB; Etanercept Psoriasis Study Group. Etanercept as monotherapy in patients with psoriasis. N Engl J Med. 2003 Nov 20;349(21):2014-22. doi: 10.1056/NEJMoa030409. PMID 14627786
- [Background] Menter A, Tyring SK, Gordon K, Kimball AB, Leonardi CL, Langley RG, Strober BE, Kaul M, Gu Y, Okun M, Papp K. Adalimumab therapy for moderate to severe psoriasis: A randomized, controlled phase III trial. J Am Acad Dermatol. 2008 Jan;58(1):106-15. doi: 10.1016/j.jaad.2007.09.010. Epub 2007 Oct 23. PMID 17936411
- [Background] Papp KA, Tyring S, Lahfa M, Prinz J, Griffiths CE, Nakanishi AM, Zitnik R, van de Kerkhof PC, Melvin L; Etanercept Psoriasis Study Group. A global phase III randomized controlled trial of etanercept in psoriasis: safety, efficacy, and effect of dose reduction. Br J Dermatol. 2005 Jun;152(6):1304-12. doi: 10.1111/j.1365-2133.2005.06688.x. PMID 15948997
- [Background] Choi SH, Chae A, Chen CH, Merki E, Shaw PX, Tsimikas S. Emerging approaches for imaging vulnerable plaques in patients. Curr Opin Biotechnol. 2007 Feb;18(1):73-82. doi: 10.1016/j.copbio.2007.01.001. Epub 2007 Jan 17. PMID 17234398
- [Background] Di Carli MF, Hachamovitch R. New technology for noninvasive evaluation of coronary artery disease. Circulation. 2007 Mar 20;115(11):1464-80. doi: 10.1161/CIRCULATIONAHA.106.629808. No abstract available. PMID 17372188
- [Background] Tardif JC, Heinonen T, Orloff D, Libby P. Vascular biomarkers and surrogates in cardiovascular disease. Circulation. 2006 Jun 27;113(25):2936-42. doi: 10.1161/CIRCULATIONAHA.105.598987. PMID 16801474
- [Background] Horiguchi J, Fujioka C, Kiguchi M, Shen Y, Althoff CE, Yamamoto H, Ito K. Soft and intermediate plaques in coronary arteries: how accurately can we measure CT attenuation using 64-MDCT? AJR Am J Roentgenol. 2007 Oct;189(4):981-8. doi: 10.2214/AJR.07.2296. PMID 17885074
- [Background] Oncel D, Oncel G, Tastan A, Tamci B. Detection of significant coronary artery stenosis with 64-section MDCT angiography. Eur J Radiol. 2007 Jun;62(3):394-405. doi: 10.1016/j.ejrad.2007.01.009. Epub 2007 Feb 15. PMID 17306490
- [Background] Pohle K, Achenbach S, Macneill B, Ropers D, Ferencik M, Moselewski F, Hoffmann U, Brady TJ, Jang IK, Daniel WG. Characterization of non-calcified coronary atherosclerotic plaque by multi-detector row CT: comparison to IVUS. Atherosclerosis. 2007 Jan;190(1):174-80. doi: 10.1016/j.atherosclerosis.2006.01.013. Epub 2006 Feb 21. PMID 16494883
- [Background] Gould KL. Positron emission tomography in coronary artery disease. Curr Opin Cardiol. 2007 Sep;22(5):422-8. doi: 10.1097/HCO.0b013e3281fc9835. PMID 17762543
- [Background] Hansson GK. Inflammation, atherosclerosis, and coronary artery disease. N Engl J Med. 2005 Apr 21;352(16):1685-95. doi: 10.1056/NEJMra043430. No abstract available. PMID 15843671
- [Derived] Bissonnette R, Tardif JC, Harel F, Pressacco J, Bolduc C, Guertin MC. Effects of the tumor necrosis factor-alpha antagonist adalimumab on arterial inflammation assessed by positron emission tomography in patients with psoriasis: results of a randomized controlled trial. Circ Cardiovasc Imaging. 2013 Jan 1;6(1):83-90. doi: 10.1161/CIRCIMAGING.112.975730. Epub 2012 Nov 30. PMID 23204039